CLINICAL TRIAL: NCT01029327
Title: Effects of Curcumin on Postprandial Blood Glucose, and Insulin in Healthy Subjects
Status: Completed | Type: Observational
Sponsor: Skane University Hospital (Other)
Other Study IDs: 353/2008c
Record Dates: First submitted 2009-12-08; First posted 2009-12-09 (Estimated); Last update posted 2009-12-09 (Estimated); Status verified 2009-06

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Healthy subjects

SUMMARY:
Previous animal studies have shown that extracts of Curcumin lowers blood glucose.

DETAILED DESCRIPTION:
To study the effect of curcumin on postprandial blood glucose and plasma concentrations of insulin in fifteen healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Fifteen healthy subjects without symptoms or a history of gastrointestinal disease, abdominal surgery or diabetes mellitus, were included in this crossover study.

Exclusion Criteria:

* Connective tissue disease or cerebrovascular or endocrine disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy subjects recruited from the population in southern Sweden.
Sampling Method: Non-Probability Sample
Dates: Start 2009-06; Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Medicine, Malmö University Hospital, Malmo, Sweden

REFERENCES:
- [Derived] Wickenberg J, Ingemansson SL, Hlebowicz J. Effects of Curcuma longa (turmeric) on postprandial plasma glucose and insulin in healthy subjects. Nutr J. 2010 Oct 12;9:43. doi: 10.1186/1475-2891-9-43. PMID 20937162